CLINICAL TRIAL: NCT01671280
Title: Drug Use Investigation Of Azithromycin Iv
Brief Title: Drug Use Investigation Of Azithromycin IV For Pneumonia Or Pelvic Inflammatory Disease (Regulatory Post Marketing Commitment Plan)
Acronym: RESCUE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0661207
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Pneumonia; Pelvic Inflammatory Disease
Keywords: pneumonia; pelvic inflammatory disease; Zithromax; Zithromac; Japanese; Regulatory Post Marketing Commitment Plan
MeSH Terms: conditions — Pneumonia; Pelvic Inflammatory Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Azithromycin IV: Subjects who are treated with Azithromycin IV
  Interventions: Drug: Azithromycin IV

INTERVENTIONS:
Drug: Azithromycin IV — The recommended dose of ZITHROMAC (azithromycin for injection) for the treatment of adult patients with pneumonia due to the indicated organisms is: 500 mg as a single daily dose by the intravenous route for at least two days. Intravenous therapy should be followed by azithromycin by the oral route at a single, daily dose of 500 mg, administered as two 250-mg tablets to complete a 7- to 10-day course of therapy.
  The recommended dose of ZITHROMAC (azithromycin for injection) for the treatment of adult patients with pelvic inflammatory disease due to the indicated organisms is: 500 mg as a single daily dose by the intravenous route for one or two days. Intravenous therapy should be followed by azithromycin by the oral route at a single, daily dose of 250 mg to complete a 7-day course of therapy.
  Other Names: Zithromac IV

SUMMARY:
To collect the efficacy and safety information of Azithromycin IV related to their appropriate use in daily practice

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients who are prescribed Zithromac IV for pneumonia or pelvic inflammatory disease.

Exclusion Criteria:

* Subjects who have been prescribed Zithromac IV for pneumonia or pelvic inflammatory disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involviong A0661207 prescribes the Zithromac IV.
Sampling Method: Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2012-09-20 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661207&StudyName=Drug%20Use%20Investigation%20Of%20Azithromycin%20IV%20For%20Community-Acquired%20Pneumonia%20Or%20Pelvic%20Inflammatory%20Disease%20%28Regulatory%20Post%20Marketing%20Commitm

RESULTS

PARTICIPANT FLOW:
Groups:
- Zithromac Intravenous Use (Azithromycin Hydrate): Participants who received Zithromac Intravenous use (and Zithromac Tablets) as indicated in the approved local product document were observed for a period of 29 days. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Started | 403 (The number is enrollment.)
Completed | 401
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: A total of 401 participants completed this study. Of the 401 participants, 1 participant was excluded from the baseline analysis due to protocol violation.
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Number analyzed (Participants) | 400
Age, Customized [Number; unit: Participants]
  <15 years | 1
  ≥15 and <65 years | 191
  ≥65 years | 208
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 194
Disease Type [Number; unit: participants] — * indicates comorbidities tabulated in duplicate.
  participants
    Pneumonia* | 299
    Pelvic inflammatory disease* | 98
    Other* | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Zithromac Intravenous use (and Zithromac Tablets) in a participant who received Zithromac Intravenous use (and Zithromac Tablets). A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to Zithromac Intravenous use (and Zithromac Tablets) was assessed by the physician.
Time Frame: 29 days
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and received Zithromac Intravenous use at least once.
Measure: Number; unit: Participants
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Number analyzed (Participants) | 400
Participants
  Treatment-Related Adverse Event | 39
  Treatment-Related Serious Adverse Event | 7

2. Secondary Outcome: Clinical Effectiveness Rate in Participants With Pneumonia
Description: Clinical effectiveness rate in participants with pneumonia, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of asssable effectiveness analysis population with pneumonia, was presented along with the corresponding 2-sided 95% CI. Clinical effectiveness of Zithromac Intravenous use (and Zithromac Tablets) was determined by the physician based on clinical symptoms and laboratory findings, and assessed according to the following categories: (1) effective, (2) ineffective, or (3) unassessable.
Time Frame: 29 days
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation of pneumonia (overall evaluation by the physician based upon change in clinical symptoms and laboratory findings) at least once. Participants evaluated as "unassessable" were excluded from the calculation.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Number analyzed (Participants) | 259
Percentage of Participants | 89.6 [85.20 to 93.02]

3. Secondary Outcome: Clinical Effectiveness Rate in Participants With Pelvic Inflammatory Disease
Description: Clinical effectiveness rate in pelvic inflammatory disease (PID), which was defined as the percentage of participants who achieved clinical effectiveness over the total number of asssable effectiveness analysis population with PID, was presented along with the corresponding 2-sided 95% CI. Clinical effectiveness of Zithromac Intravenous use (and Zithromac Tablets) was determined by the physician based on clinical symptoms and laboratory findings, and assessed according to the following categories: (1) effective, (2) ineffective, or (3) unassessable.
Time Frame: 29 days
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation of PID (overall evaluation by the physician based upon change in clinical symptoms and laboratory findings) at least once. Participants evaluated as "unassessable" were excluded from the calculation.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Number analyzed (Participants) | 91
Percentage of Participants | 91.2 [83.41 to 96.13]

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Zithromac Intravenous Use (Azithromycin Hydrate)
Serious Adverse Events (participants affected / at risk) | 43/400
Other Adverse Events (participants affected / at risk) | 34/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zithromac Intravenous Use (Azithromycin Hydrate) (N=400)
Clostridium difficile colitis (Infections and infestations) | 1
Gastroenteritis staphylococcal (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 12
Peritonitis (Infections and infestations) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 3
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zithromac Intravenous Use (Azithromycin Hydrate) (N=400)
Insomnia (Psychiatric disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 14
Hepatic function abnormal (Hepatobiliary disorders) | 9
Liver disorder (Hepatobiliary disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.